CLINICAL TRIAL: NCT05249465
Title: Optimizing Self-monitoring in a Digital Health Intervention for Weight Loss
Brief Title: Spark: Finding the Optimal Tracking Strategy for Weight Loss in a Digital Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michele Patel, Instructor, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 64716; K23DK129805 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Overweight; Weight Loss; Health Behavior
Keywords: digital health; mobile health; intervention; weight loss; behavioral treatment; Multiphase Optimization Strategy (MOST); obesity treatment; dietary change; physical activity; self-monitoring; factorial design
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study uses a full factorial experimental design testing the efficacy of three intervention components, each with two levels (i.e., a 2x2x2).
Masking Description: Outcomes will be analyzed in a blinded fashion such that treatment allocation is not revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): Core Only
  Interventions: Behavioral: Core behavioral weight loss intervention
- Condition 2 (Experimental): Core + Track Weight
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring weight
- Condition 3 (Experimental): Core + Track Steps
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring steps
- Condition 4 (Experimental): Core + Track Diet
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring diet
- Condition 5 (Experimental): Core + Track Weight + Track Steps
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring weight; Behavioral: Self-monitoring steps
- Condition 6 (Experimental): Core + Track Weight + Track Diet
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring diet; Behavioral: Self-monitoring weight
- Condition 7 (Experimental): Core + Track Steps + Track Diet
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring diet; Behavioral: Self-monitoring steps
- Condition 8 (Experimental): Core + Track Weight + Track Steps + Track Diet
  Interventions: Behavioral: Core behavioral weight loss intervention; Behavioral: Self-monitoring diet; Behavioral: Self-monitoring weight; Behavioral: Self-monitoring steps

INTERVENTIONS:
Behavioral: Core behavioral weight loss intervention — All participants will receive a 6-month "core" behavioral obesity treatment consisting of goal setting, behavioral lessons, action plans, and tailored feedback - all of which will be delivered remotely.
Behavioral: Self-monitoring diet — Participants randomized to receive this component will be instructed to self-monitor their dietary intake daily via the Fitbit mobile app. Participants will receive a daily calorie goal.
  Arms: Condition 4; Condition 6; Condition 7; Condition 8
Behavioral: Self-monitoring weight — Participants randomized to receive this component will be instructed to self-monitor their body weight daily via a wireless e-scale (e.g., the Fitbit Aria Scale).
  Arms: Condition 2; Condition 5; Condition 6; Condition 8
Behavioral: Self-monitoring steps — Participants randomized to receive this component will be instructed to self-monitor their step count daily via a wrist-worn Fitbit activity monitor. A daily step goal will be given that will adapt based on progress.
  Arms: Condition 3; Condition 5; Condition 7; Condition 8

SUMMARY:
This optimization trial will examine three tracking (or "self-monitoring") strategies for weight loss -- tracking dietary intake, steps, and/or body weight -- all delivered through digital health tools. The purpose of the study is to evaluate the combination of these strategies that maximizes 6-month weight loss in the context of a standalone digital health intervention for adults with overweight or obesity.

The investigators will recruit 176 total participants to the trial. Recruitment will occur through remote channels. Interested individuals will be directed to an online screening questionnaire; those who are eligible will then be invited to attend an initial remote session with study personnel to ensure interest and eligibility in the study. The weight loss intervention will last 6 months, and all participants will receive a "core" treatment consisting of goal setting, behavioral lessons, action plans, and tailored feedback - all of which will be delivered remotely. Depending on which group participants are assigned to in the study, some individuals will be asked to track their dietary intake, their steps, and/or their body weight via digital tools. All study tasks will occur remotely, thus, participants never need to come in-person for any intervention or assessment tasks.

The investigators will use the Multiphase Optimization Strategy (MOST) framework to identify the most effective combination of self-monitoring strategies. The factorial design will allow the research team to determine the unique and combined impact of each self-monitoring component on weight change. The primary outcome is weight change from baseline to 6 months. The research team will also assess self-monitoring engagement over 6 months and its association with weight change. To complement the main trial, the research team will also randomize half of participants to receive an interactive orientation video, in order to assess its impact on trial retention at 6 months. Overall, the information gathered from this trial will enable the construction of an optimized digital health intervention for weight loss that can be delivered remotely, which, if found to be effective, could have high potential for scalability.

ELIGIBILITY:
Inclusion Criteria:

* adults (ages 18+ years)
* body mass index (BMI) 25.0 to 45.0 kg/m^2
* smartphone ownership
* willingness to install a mobile app on their phone
* access to a personal email account
* English language proficiency
* interest in losing weight through behavioral strategies

Exclusion Criteria:

* concurrent enrollment in another weight management intervention
* loss of ≥10 lbs. in the past 6 months
* current use of a weight loss medication
* prior or planned bariatric surgery
* current or planned pregnancy in the trial period
* currently breastfeeding
* lives with someone else participating in the study
* hospitalization for a mental health condition in the past 12 months
* inability to engage in moderate forms of physical activity akin to brisk walking (assessed by the Physical Activity Readiness Questionnaire)
* if weight loss is contraindicated or might be impacted by a condition or medication (e.g., end stage renal disease, cancer, schizophrenia, dementia, steroids, anti-psychotics)
* if an individual would be better suited for a more intensive or different type of intervention based on a health condition (e.g., individuals with history of an eating disorder or cardiovascular event, uncontrolled hypertension, or uncontrolled diabetes mellitus)
* investigator discretion for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Body weight change from baseline to 6 months | baseline, 6 months
  change in weight from baseline to 6-month followup (in kg); assessed objectively via e-scale

SECONDARY OUTCOMES:
Body weight from baseline to 1 month | baseline, 1 month
  change in weight from baseline to 1-month followup (in kg); assessed objectively via e-scale
Body weight from baseline to 3 months | baseline, 3 month
  change in weight from baseline to 3-month followup (in kg); assessed objectively via e-scale
Clinically significant weight loss | 6 months
  proportion of participants achieving ≥5% weight loss from baseline
BMI change from baseline to 6 months | baseline, 6 months
  change in BMI from baseline to 6-month followup (in kg/m^2); computed from self-reported height and e-scale weight
Caloric intake change from baseline to 6 months | baseline, 6 months
  change in caloric intake from baseline to 6-month followup (in kcal); assessed using Automated 24-Hour (ASA-24) Dietary Assessment Tool (2 separate 24hr diet recalls at each time point: 1 week day, 1 weekend day)
Physical activity change from baseline to 6 months | baseline, 6 months
  change in physical activity from baseline to 6-month followup; assessed using Godin Leisure-Time Exercise Questionnaire
Engagement in self-monitoring dietary intake | 6 months of the intervention
  average percent of days in the 6-month intervention of self-monitoring dietary intake; assessed objectively via digital health tools (mobile app)
Engagement in self-monitoring weight | 6 months of the intervention
  average percent of days in the 6-month intervention of self-monitoring weight; assessed objectively via digital health tools (e-scale)
Engagement in self-monitoring steps | 6 months of the intervention
  average percent of days in the 6-month intervention of self-monitoring steps; assessed objectively via digital health tools (activity monitor)

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Patel, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Once the study data have undergone final data cleaning, analysis, and planned publications, the investigators will make the final data collected as part of the proposed research available in electronic form to researchers who request them. Researchers will be asked to submit a data request in writing to the Principal Investigator so that the requested data can be made available while protecting the confidentiality of study participants and ensuring that the proposed research questions do not overlap with planned publication development by the project research team or other groups. The requested dataset will be free of identifiers that would permit linkages to individual research participants. The requestor must agree to maintain the privacy and confidentiality of the data and must indicate how they plan to store the data to demonstrate compliance with secure computing. All publications that emerge from this award will be publicly available via PubMed Central.

REFERENCES:
- [Derived] Patel ML, King AC, Rosas LG, Bennett GG, Collins LM, Gallis JA, Zeitlin AB, Talreja PS, Crosthwaite PC, Collins KA, Lim AW, Kim TS. Optimizing Self-Monitoring in a Digital Weight Loss Intervention (Spark): Protocol for a Factorial Randomized Trial. JMIR Res Protoc. 2025 Sep 23;14:e75629. doi: 10.2196/75629. PMID 40986860

DOCUMENTS (2):
  • Study Protocol (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05249465/Prot_000.pdf
  • Informed Consent Form (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT05249465/ICF_001.pdf